CLINICAL TRIAL: NCT01819935
Title: Clinical Outcomes Among a National Veterans Affairs Methicillin Resistant Staphylococcus Aureus (MRSA) Pneumonia Cohort Treated With Linezolid Or Vancomycin
Brief Title: Clinical Outcomes of Methicillin Resistant Staphylococcus Aureus (MRSA) Hospital-Based Pneumonia
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5951163
Record Dates: First submitted 2013-02-28; First posted 2013-03-28 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-12

CONDITIONS: Pneumonia
Keywords: MRSA. pneumonia; outcomes
MeSH Terms: conditions — Pneumonia | interventions — Linezolid; Vancomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- linezolid (Zyvox)
  Interventions: Drug: linezolid (Zyvox)
- Vancomycin
  Interventions: Drug: vancomycin

INTERVENTIONS:
Drug: linezolid (Zyvox) — As prescribed-this is retrospective cohort of existing clinical data.
  Groups: linezolid (Zyvox)
Drug: vancomycin — As prescribed-this is retrospective cohort of existing clinical data.
  Groups: Vancomycin

SUMMARY:
The purpose of this non-interventional, retrospective study of existing data is to evaluate clinical outcomes related to Methicillin-resistant Staphylococcus aureus hospital based pneumonia by treatment and among subpopulations.

DETAILED DESCRIPTION:
All patients meeting inclusion/exclusion criteria from inpatient database from 1/1/02-9/30/10.

ELIGIBILITY:
Inclusion Criteria:

* MRSA and pneumonia cases by ICD-9 code identification.
* Diagnosis included during inpatient stay.
* Treatment initiation in hospital.

Exclusion Criteria:

* Death of discharge within 3 days of treatment initiation.
* Exposure to other treatments with MRSA activity.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: National database of inpatient admissions between January 1, 2002 and Septmeber 30, 2010
Sampling Method: Non-Probability Sample
Enrollment: 5271 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951163&StudyName=Clinical%20Outcomes%20of%20Methicillin%20Resistant%20Staphylococcus%20Aureus%20%28MRSA%29%20Hospital-Based%20Pneumonia

RESULTS

PARTICIPANT FLOW:
Groups:
- Linezolid: Participants who were admitted to veterans affairs hospitals between 1 January 2001 and 30 September 2010 (3559 days) with an international classification of diseases - revision 9 (ICD-9) code for methicillin-resistant staphylococcus aureus (MRSA) and pneumonia, who had initiated and received at least 3 days of continuous intravenous or oral linezolid therapy in the hospital, were analyzed retrospectively.
- Vancomycin: Participants who were admitted to veterans affairs hospitals between 1 January 2001 and 30 September 2010 (3559 days) with an ICD-9 code for MRSA and pneumonia, who had initiated and received at least 3 days of continuous intravenous vancomycin therapy in the hospital, were analyzed retrospectively.
Period: Overall Study
Arm/Group | Linezolid | Vancomycin
Started | 328 | 4943
Completed | 328 | 4943
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were admitted to veterans affairs hospitals between 1 January 2001 and 30 September 2010 (3559 days) with an ICD-9 code for MRSA and pneumonia.
Groups:
- Total: Total of all reporting groups
Arm/Group | Linezolid | Vancomycin | Total
Number analyzed (Participants) | 328 | 4943 | 5271
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (12.5) | 69.1 (12.7) | 69.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 99 | 104
  Male | 323 | 4844 | 5167

OUTCOME MEASURES:

1. Primary Outcome: Time to 30-day Mortality
Description: Time to death (all-cause mortality) occurring within 30 days of treatment initiation was reported. Mortality was assessed from admission vital status databases.
Time Frame: Baseline (1 January 2001) up to 3559 Days (30 September 2010)
Population: FAS included all participants who were admitted to veterans affairs hospitals between 1 January 2001 and 30 September 2010 (3559 days) with an ICD-9 code for MRSA and pneumonia.
Measure: Median (Full Range); unit: days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 328 | 4943
days | 15 [3 to 30] | 14 [3 to 30]
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Propensity Cox proportional hazards regression model was used; Test type: Superiority or Other; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.72 to 1.20]

2. Secondary Outcome: Time to Therapy Change
Description: Time to therapy change was calculated from initiation of therapy (index date) to change in therapy (event date). Therapy change was defined as the discontinuation of linezolid or vancomycin and initiation of a different agent with activity against MRSA (clindamycin, daptomycin, doxycycline, linezolid, minocycline, tigecycline, trimethoprim/sulfamethoxazole, vancomycin). As such, therapy change included switching from linezolid to vancomycin, switching from vancomycin to linezolid, or switching from either linezolid or vancomycin to another anti-MRSA antibiotic.
Time Frame: Baseline (1 January 2001) up to 3559 Days (30 September 2010)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 328 | 4943
days | 4 [3 to 6] | 4 [3 to 7]
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Propensity Cox proportional hazards regression model was used; Test type: Superiority or Other; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.53 to 1.05]

3. Secondary Outcome: Time to Discharge From the Hospital
Description: Time to discharge from hospital was calculated from initiation of therapy (index date) to hospital discharge (event date).
Time Frame: Baseline (1 January 2001) up to 3559 Days (30 September 2010)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 328 | 4943
days | 19.7 (24.4) | 20.3 (26.5)
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Propensity Cox proportional hazards regression model was used; Test type: Superiority or Other; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.90 to 1.15]

4. Secondary Outcome: Time to Transfer Out From the Intensive Care Unit (ICU)
Description: Time to discharge from the ICU was calculated from the initiation of therapy (index date) to the time the participant was transferred out from ICU (event date). Transfer out of an ICU was assessed among those participants who had initiated linezolid or vancomycin therapy in the ICU.
Time Frame: Baseline (1 January 2001) up to 3559 Days (30 September 2010)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 328 | 4943
days | 2 [1 to 14] | 4 [1 to 14]
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Propensity Cox proportional hazards regression model was used; Test type: Superiority or Other; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.39 to 1.09]

5. Secondary Outcome: Time to Intubation
Description: Time to intubation was calculated from the initiation of therapy (index date) to intubation (event date).
Time Frame: Baseline (1 January 2001) up to 3559 Days (30 September 2010)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 328 | 4943
days | 5 [1 to 59] | 3 [1 to 28]
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Propensity Cox proportional hazards regression model was used; Test type: Superiority or Other; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.68 to 1.37]

6. Secondary Outcome: Time to 30-day Re-admission
Description: Time to readmission to any veterans affairs hospital facility within 30 days after hospital discharge was reported.
Time Frame: Baseline (1 January 2001) up to 3559 Days (30 September 2010)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 328 | 4943
days | 10 [1 to 30] | 11 [1 to 30]
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Propensity Cox proportional hazards regression model was used; Test type: Superiority or Other; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.68 to 1.13]

7. Secondary Outcome: Time to 30-day Methicillin-Resistant Staphylococcus Aureus (MRSA) Re-infection
Description: Time to MRSA re-infection was defined as readmission with MRSA infection to any veterans affairs hospital facility within 30 days after hospital discharge.
Time Frame: Baseline (1 January 2001) up to 3559 Days (30 September 2010)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 328 | 4943
days | 17 [2 to 30] | 11 [1 to 30]
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Propensity Cox proportional hazards regression model was used; Test type: Superiority or Other; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.54 to 1.48]

8. Secondary Outcome: Clinical Success
Description: Clinical success, a composite outcome defined as discharge from the hospital or ICU by day 14 after treatment initiation, in the absence of death, therapy change, or intubation by day 14. Percentage of participants with clinical success was reported.
Time Frame: Baseline (1 January 2001) up to 3559 Days (30 September 2010)
Population: FAS included all participants who were admitted to veterans affairs hospitals between 1 January 2001 and 30 September 2010 (3559 days) with an ICD-9 code for MRSA and pneumonia. Here, "N" (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 231 | 3500
percentage of participants | 50.9 | 46
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Propensity Cox proportional hazards regression model was used; Test type: Superiority or Other; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [1.06 to 1.45]

ADVERSE EVENTS:
Description: This retrospective study used participants-level electronic health related databases (e-HRD), in which it was not possible to link (i.e. identify a potential association between) a particular product and medical event for any individual. Thus, adverse events (AEs) were not reportable as individual AE reports.
Arm/Group | Linezolid | Vancomycin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Results for 'time to intubation' was reported and not 'time to extubation' due to change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.